CLINICAL TRIAL: NCT02236676
Title: Sleep, Procedural Learning & Therapeutic Engagement Among Inpatients With
Brief Title: Sleep Study Among Inpatients With TBI in an Acute Rehabilitation Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Principal Investigator, Anthony Lequerica, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-833-14
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Motor Learning in TBI
Keywords: motor learning TBI

ARMS (2):
- Nap after rehearsal trials (Active Comparator): A 30-minute daytime nap after training
  Interventions: Behavioral: Nap after rehearsal trials
- Resting while awake (Placebo Comparator): Placebo condition of 30 minutes between training and retesting in which the half hour is spent resting awake in bed.
  Interventions: Behavioral: Nap after rehearsal trials

INTERVENTIONS:
Behavioral: Nap after rehearsal trials — Behavioral

SUMMARY:
The purpose of this research study is to better understand how a daytime nap after training on a motor skill after brain injury improves performance compared with the same amount of time after training spent awake and resting.

ELIGIBILITY:
Inclusion Criteria:

* Must have a Traumatic Brain Injury.
* Must have been a Kessler Institute for Rehabilitation inpatient for at least three days.

Exclusion Criteria:

* Bilateral arm fractures, cellulitis or other conditions that prevent safe wearing of the WatchPAT-200/actigragh.
* Movement disorder or spasticity affecting both upper extremities
* Patients who are ventilator-dependent.
* Patients who are on contact precautions for C.diff or other highly contagious diseases.
* Patients with neurological disorders other than TBI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement on Motor Functioning Test | Three Nights and Three Days
  Change scores from day 1 to day 3 will be compared in both Nap and No Nap conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States